CLINICAL TRIAL: NCT01361958
Title: Double-blind, Comparative, Randomized, Single Center, Between-subject, Dose-finding Clinical Trial to Compare 4 Doses of the Combination 17beta-estradiol/Nomegestrol Acetate Administered From Day 1 to Day 21 of the Menstrual Cycle on the Inhibition of Ovulation
Brief Title: Minimal Effective Dose of Nomegestrol Acetate Inhibiting the Ovulation in Women Receiving Estradiol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theramex (Industry)
Responsible Party: Dr Didier Chassard, Aster, Paris, France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96-ESC/NOM-1-RD
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Suppression of Ovulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- T1 received 0.625 mg NOMAC + 1.5 mg E2 (Experimental)
  Interventions: Drug: NOMAC
- T2 received 1.25 mg NOMAC + 1.5 mg E2 (Experimental)
  Interventions: Drug: NOMAC
- T3 received 2.5 mg NOMAC + 1.5 mg E2 (Experimental)
  Interventions: Drug: NOMAC
- T4 received 2.5 mg NOMAC + Lactose (Experimental)
  Interventions: Drug: NOMAC

INTERVENTIONS:
Drug: NOMAC

SUMMARY:
The aim of the present study was to evaluate the ability of several doses of NOMAC in combination with E2 to inhibit ovulation and to assess changes in the gonadotropin and ovarian hormone profiles, in comparison to a control cycle in healthy-volunteer premenopausal women.

The study was also designed to check whether the combined administration of E2 and NOMAC at the dose of 2.5 mg daily induces any changes in the effects of the progestin compared to when it is given alone.

ELIGIBILITY:
Inclusion Criteria:

* Female premenopausal healthy volunteers having given their informed written consent at the first selection visit,
* Registered with Social Security in agreement with the French Law on biomedical research on volunteers,
* Sufficiently co-operative to meet the needs of the study,
* Accepting not to become pregnant during the trial,
* Accepting the use of condoms as the single authorized contraceptive means during the trial,
* With a diurnal and regular job or activity,
* Aged 18 to 35 years old inclusive,
* Non-smokers or current smokers of less than 10 cigarettes/day,
* With normal eating habits,
* With a body mass index between 17 and 27 inclusive,

Exclusion Criteria:

* Participation in another clinical trial,
* Blood donation in the three months prior to Visit V1 or intention to donate blood during the trial or within the three months following the trial completion,
* Virgins, because of the gynecological examination,
* Subjects who were within the exclusion period in the Healthy Volunteers National Register of the French Ministry of Health,
* Forfeiture of freedom by administrative or legal award or under guardianship,
* No possible contact in case of emergency,
* Strenuous physical activity planned during the trial. Concerning the gynecological status and examination
* History of major medical, psychiatric illness or surgery,
* Any acute or chronic systemic disease or disorder,
* History of hypersensitivity to at least one drug (abnormal drug reaction or idiosyncrasy or asthma),
* Abuse of alcohol i.e. history or evidence of acute or chronic abuse, more than 45 g of alcohol per day,
* Excessive drinking of tea, coffee, chocolate, and/or beverages containing caffeine (>5 cups/day or approximately 500 mg of caffeine per day),
* Current vascular pathology or with a past history of thrombo-embolic disease, arterial hypertension (BPS ≥ 160 mm Hg or BPD ≥ 95 mm Hg), coronary artery disease, valvulopathy; thrombogenic cardiac rhythm disturbances, cerebrovascular disease, ocular pathology of vascular origin,
* Cancer or progressive hematological disorder,
* Current or past history of pituitary tumors,
* Epilepsy,
* Known hyperprolactinemia,
* Known renal insufficiency,
* Severe or recent liver disease or symptomatic vesicular lithiasis, or recurrent cholestasis or recurring pruritus of pregnancy,
* Abnormality (> 1N) in liver function on the selection laboratory investigation (ALT or AST > 50 IU/L or alkaline phosphatases > 125 IU/L or total bilirubin > 22 μmol/L or GGT > 70 IU/L),
* Known diabetes or fasting blood sugar > 6.2 mmol/L (1N) at the selection laboratory investigation,
* Uncontrolled treated dyslipidemia or cholesterolemia > 5.2 mmol/L (93%N), then > 6.2 mmol/L (110%N) after protocol amendment during the course of the study, or triglyceridemia > 1.80 mmol/L (79 %N) at the selection laboratory investigation,
* Plasma creatinine > 115 μmol/L (1N),
* Abnormality in any of the hematology parameters,
* Positive results at any of the serologies (HBs antigen, HCV antibodies, HIV 1 & 2 antibodies) performed at V1,
* Positive result for β-HCG at any measurements (i.e. β-HCG > 5 mIU/mL),
* Abnormality in the baseline EKG,
* Connective tissue disorder,
* Porphyria,
* Otosclerosis,
* Abnormality at the medical examination performed at V1 which included a neurological examination,
* Past history or clinical evidence of any malignant tumor or benign disease of the breasts or uterus or ovary (including endometriosis, leiomyomas, polycystic ovaries ...),
* Vaginal infection at the vaginal bacteriological examination performed at V1. After protocol amendment during the course of the study, infection diagnosed at the vaginal bacteriology or at the cervico-vaginal smear was removed from the exclusion criteria list.
* Hysterectomy, even partial, or endometrectomy,
* Pregnancy,
* Childbirth, breast-feeding, miscarriage or termination of pregnancy in the year prior to V1,

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 1997-02; Primary Completion 1997-11 (Actual); Study Completion 1998-09 (Actual)